CLINICAL TRIAL: NCT00857506
Title: Longitudinal Study of Long-term (36 Month) Cognitive Outcomes in Healthy Volunteers, Patients With Mild Cognitive Impairment (MCI) and Patients With Alzheimer's Disease (AD) Who Have Previously Had PET Imaging With 18F-AV-45 Injection.
Brief Title: Observational Study of Cognitive Outcomes for Subjects Who Have Had Prior PET Amyloid Imaging With Florbetapir F 18 (18F-AV-45)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18F-AV-45-A11
Record Dates: First submitted 2009-03-05; First posted 2009-03-06 (Estimated); Results first posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
Keywords: Cognitive outcome; 18F-AV-45 PET scan; Amyloid PET scan; Florbetapir F 18 amyloid PET scan; Normal cognition; Change in cognitive status in relation to brain amyloid on PET
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — florbetapir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: florbetapir F 18 — 370 Mega Becquerel (10 mCi)
  Other Names: 18F-AV-45 PET; amyloid imaging; Amyvid

SUMMARY:
The primary objective of this protocol is to determine if brain amyloid imaged with florbetapir F 18 (18F-AV-45) PET scans is predictive of progressive cognitive impairment during the subsequent 36 months for groups of: normal controls, mild cognitive impairment and Alzheimer's disease.

Hypothesis 1: The probability a subject will experience progressive cognitive impairment within 36 months of imaging will be greater in subjects whose 18F-AV-45 PET scan was rated amyloid positive compared to subjects whose PET scan was rated amyloid negative.

The secondary objective is to determine the stability, over 36 months of a clinical diagnosis, of AD in patients with an amyloid positive 18F-AV-45 PET.

Hypothesis 2: The diagnosis of AD will remain unchanged in patients whose PET scan were rated as amyloid positive.

DETAILED DESCRIPTION:
Study AV-45-A11 is designed to determine if brain amyloid aggregation imaged on 18F-AV-45 PET scans is predictive of progression of cognitive impairment during the subsequent 36 months. Approximately 180 subjects enrolled in a prior clinical study (AV-45-A05[NCT00702143]) will be offered an opportunity to be studied under this protocol. The initial visit will occur as soon as possible following the AV-45-A05(NCT00702143) imaging day. Subjects who qualify for the study and their caregiver/partners will be contacted approximately 6,12,18,24 and 36 months after PET imaging in study AV-45-A05(NCT00702143), and will undergo a standardized functional and psychometric evaluation.

NOTE: This study is a clinical follow-up of subjects previously enrolled in trial 18F-AV-45-A05(NCT00702143). No new patients are being enrolled in this trial.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who enrolled in study AV-45-A05(NCT00702143), received 18F-AV-45, and completed a PET scan will be eligible to enroll in this trial.

Exclusion Criteria:

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (8):
- United States (8):
  - Research Site, Scottsdale, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Costa Mesa, California
  - Research Site, Brooksville, Florida
  - Research Site, Hallandale, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Albany, New York
  - Research Site, Durham, North Carolina

REFERENCES:
- [Derived] Siderowf A, Pontecorvo MJ, Shill HA, Mintun MA, Arora A, Joshi AD, Lu M, Adler CH, Galasko D, Liebsack C, Skovronsky DM, Sabbagh MN. PET imaging of amyloid with Florbetapir F 18 and PET imaging of dopamine degeneration with 18F-AV-133 (florbenazine) in patients with Alzheimer's disease and Lewy body disorders. BMC Neurol. 2014 Apr 9;14:79. doi: 10.1186/1471-2377-14-79. PMID 24716655

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from participants in study 18F-AV-45-A05 (NCT00702143)
Groups:
- Alzheimer's Disease: Subject's with Alzheimer's Disease were recruited from study 18F-AV-45-A05 (NCT00702143). None of these subjects received additional interventions in study 18F-AV-45-A11.
- Mild Cognitive Impairment: Subject's with Mild Cognitive Impairment (MCI) were recruited from study 18F-AV-45-A05 (NCT00702143). 36 of these subjects received a single dose of florbetapir F 18 370 MBq (10 mCi), IV injection at the 24 month time point of study 18F-AV-45-A11 and comprise the safety set discussed in the Adverse Events section.
- Cognitively Normal: Cognitively Normal (CN) subjects were recruited from study 18F-AV-45-A05 (NCT00702143). 50 of these subjects received a single dose of florbetapir F 18 370 MBq (10 mCi), IV injection at the 24 month time point of study 18F-AV-45-A11 and comprise the safety set discussed in the Adverse Events section.
Period: Overall Study
Arm/Group | Alzheimer's Disease | Mild Cognitive Impairment | Cognitively Normal
Started | 31 | 52 | 69
Completed | 16 | 37 | 51
Not Completed | 15 | 15 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alzheimer's Disease | Mild Cognitive Impairment | Cognitively Normal | Total
Number analyzed (Participants) | 31 | 52 | 69 | 152
Age Continuous [Mean (Standard Deviation); unit: years] | 76.7 (9.23) | 71.5 (10.09) | 69.8 (11.26) | 71.8 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 29 | 41 | 83
  Male | 18 | 23 | 28 | 69
Region of Enrollment [Number; unit: participants]
  United States | 31 | 52 | 69 | 152

OUTCOME MEASURES:

1. Primary Outcome: Change in ADAS-Cog for MCI Subjects
Description: The primary analysis was the comparison in the magnitude of change from baseline in Alzheimer's Disease Assessment Scale cognitive subscale (ADAS-Cog) between Aβ+ and Aβ- subjects in the Mild Cognitive Impairment (MCI) population at 36 months adjusting for baseline test score and age at informed consent. ADAS-Cog scores (range 0-70) indicate performance on a series of 11 cognitive tasks where 0 indicates the highest level of cognitive performance and 70 indicates the lowest level of cognitive performance. Change in ADAS-Cog scores were calculated by subtracting the baseline score from the 36 month score (last observation carried forward [LOCF]). A change in ADAS-Cog greater than 0 indicates a deterioration in cognitive performance whereas a change in ADAS-Cog less than 0 indicates improved cognitive performance.
Time Frame: Baseline and 36 months
Population: Brain amyloid status was determined by baseline florbetapir F 18 PET scans performed in study 18F-AV-45-A05 (NCT00702143).
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Amyloid-Beta Positive MCI Subjects: MCI subjects with a positive florbetapir F 18 PET scan at baseline.
- Amyloid-Beta Negative MCI Subjects: MCI subjects with a negative florbetapir F 18 PET scan at baseline.
Arm/Group | Amyloid-Beta Positive MCI Subjects | Amyloid-Beta Negative MCI Subjects
Number analyzed (Participants) | 17 | 30
Scores on a scale | 5.664 (1.4667) | -0.710 (1.0905)

2. Secondary Outcome: Cognitive Decline in MCI Subjects
Description: The key secondary analyses compared the number of Aβ+ and Aβ- subjects in the MCI population with clinically significant deterioration in ADAS-Cog (≥4) and Clinical Dementia Rating (CDR) global score (≥0.5) and conversion in diagnosis from MCI at baseline to AD or Cognitively Normal (CN) at 36 months. ADAS-Cog scores (range 0-70) indicate performance on a series of 11 cognitive tasks where 0 indicates the highest level of cognitive performance and 70 indicates the lowest level of cognitive performance. CDR scores (range 0-3) quantify the severity of the symptoms of dementia where 0 indicates no cognitive impairment and 3 indicates severe dementia. Changes in ADAS-Cog and CDR scores were calculated by subtracting the baseline score from the 36 month score (LOCF).
Time Frame: Baseline and 36 months
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Amyloid-Beta Positive MCI Subjects | Amyloid-Beta Negative MCI Subjects
Number analyzed (Participants) | 17 | 30
Participants
  ADAS-Cog Deterioration ≥4 | 8 | 3
  CDR Deterioration ≥0.5 | 5 | 4
  Conversion to AD | 6 | 3
  Conversion to CN | 1 | 5

3. Secondary Outcome: Change in ADAS-Cog in CN and AD Subjects
Description: This analysis compared the magnitude of change from baseline in ADAS cognitive subscale (ADAS-Cog) scores between Aβ+ and Aβ- subjects in the CN and AD populations at 36 months adjusting for baseline test score and age at informed consent. ADAS-Cog scores (range 0-70) indicate performance on a series of 11 cognitive tasks where 0 indicates the highest level of cognitive performance and 70 indicates the lowest level of cognitive performance. Change in ADAS-Cog scores were calculated by subtracting the baseline score from the 36 month score (LOCF). A change in ADAS-Cog greater than 0 indicates a deterioration in cognitive performance whereas a change in ADAS-Cog less than 0 indicates improved cognitive performance.
Time Frame: Baseline and 36 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Amyloid-Beta Positive CN Subjects: CN subjects with a positive florbetapir F 18 PET scan at baseline.
- Amyloid-Beta Negative CN Subjects: CN subjects with a negative florbetapir F 18 PET scan at baseline.
- Amyloid-Beta Positive AD Subjects: AD subjects with a positive florbetapir F 18 PET scan at baseline.
- Amyloid-Beta Negative AD Subjects: AD subjects with a negative florbetapir F 18 PET scan at baseline.
Arm/Group | Amyloid-Beta Positive CN Subjects | Amyloid-Beta Negative CN Subjects | Amyloid-Beta Positive AD Subjects | Amyloid-Beta Negative AD Subjects
Number analyzed (Participants) | 10 | 57 | 19 | 9
Scores on a scale | 3.237 (0.9043) | -0.094 (0.3679) | 8.879 (2.8812) | 3.811 (4.4261)

4. Secondary Outcome: Cognitive Decline in CN and AD Subjects
Description: The key secondary analyses compared the number of Aβ+ and Aβ- subjects in the CN and AD populations with clinically significant deterioration in ADAS-Cog (≥4) and CDR global score (≥0.5). ADAS-Cog scores (range 0-70) indicate performance on a series of cognitive tasks where 0 indicates the highest level of cognitive performance and 70 indicates the lowest level of cognitive performance. CDR scores (range 0-3) quantify the severity of the symptoms of dementia where 0 indicates no cognitive impairment and 3 indicates severe dementia. Changes in ADAS-Cog and CDR scores were calculated by subtracting the baseline score from the 36 month score (LOCF).
Time Frame: Baseline and 36 months
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- Amyloid-Beta Negative CN Subjects: CN subjects with a negative florbetapir F 18 PET scan at baseline. 57 subjects were analyzed for change in ADAS-Cog and 55 subjects were analyzed for change in CDR.
Arm/Group | Amyloid-Beta Positive CN Subjects | Amyloid-Beta Negative CN Subjects | Amyloid-Beta Positive AD Subjects | Amyloid-Beta Negative AD Subjects
Number analyzed (Participants) | 10 | 57 | 19 | 9
Participants
  ADAS-Cog Deterioration ≥4 | 4 | 3 | 14 | 3
  CDR Deterioration ≥0.5 | 4 | 5 | 12 | 2

5. Secondary Outcome: Covariate Adjusted Psychometric Score Change
Description: Change from baseline by diagnostic group in covariate-adjusted psychometric assessment scores at month 36 (LOCF). Assessments included Digit Symbol Substitution (DSS), Clinical Dementia Rating Sum of Boxes (CDR-SOB), Mini-Mental State Examination (MMSE), Wechsler Logical Memory Scale (WLMS) delayed and immediate recall, Category Verbal Fluency (CVF) animals and vegetables, Alzheimer's Disease Clinical Studies Consortium Activities of Daily Living (ADCS ADL) and Geriatric Depression Scale (GDS). The ranges for these scales are as follows: DSS (0-93), CDR-SOB (0-18), MMSE (0-30), WLMS delayed and immediate recall (0-25), CVF animals and vegetables (0-total number of relevant items named in 60 seconds), ADCS ADL (0-78) and GDS (0-15). For all scales except CDR-SOB and GDS a higher score indicates greater cognitive function. For CDR-SOB and GDS a higher score indicates increased dementia or depression, respectively.
Time Frame: Baseline and 36 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale
Groups:
- Amyloid-Beta Negative CN Subjects: CN subjects with a negative florbetapir F 18 PET scan at baseline. All assessments were obtained for 57 subjects except for CDR-SOB and ADCS ADL which were obtained for 55 and 56 subjects respectively.
Arm/Group | Amyloid-Beta Positive CN Subjects | Amyloid-Beta Negative CN Subjects | Amyloid-Beta Positive MCI Subjects | Amyloid-Beta Negative MCI Subjects | Amyloid-Beta Positive AD Subjects | Amyloid-Beta Negative AD Subjects
Number analyzed (Participants) | 10 | 57 | 17 | 30 | 19 | 9
Scores on a scale
  DSS | -6.521 (2.9117) | 0.214 (1.1709) | -10.940 (2.1569) | 0.133 (1.6082) | -5.995 (2.2381) | -0.011 (3.3534)
  CDR-SOB | 0.765 (0.1520) | 0.097 (0.0632) | 1.985 (0.5321) | 0.392 (0.3976) | 4.048 (0.8008) | 0.121 (1.1739)
  MMSE | -0.740 (0.3282) | -0.396 (0.1329) | -2.882 (0.8053) | -0.300 (0.6023) | -3.924 (1.2418) | 1.173 (1.8299)
  WLMS delayed recall | -0.429 (1.1278) | 0.970 (0.4504) | -1.459 (1.1250) | 0.493 (0.8386) | -0.179 (0.6722) | 1.490 (1.10058)
  WLMS immediate recall | -0.926 (1.0560) | 0.934 (0.4211) | -1.875 (0.9949) | 0.496 (0.7405) | -0.891 (0.8151) | -0.231 (1.2620)
  CVF animals | -2.785 (1.5735) | -0.617 (0.6383) | -3.177 (1.0980) | -0.533 (0.8213) | -4.772 (0.8096) | 0.085 (1.2654)
  CVF vegetables | -2.087 (1.0202) | 0.156 (0.4150) | -2.278 (0.8162) | 0.757 (0.6109) | -3.051 (0.7022) | 0.621 (1.0959)
  ADCS ADL | -0.629 (0.7272) | -0.191 (0.2796) | -4.932 (2.2040) | -2.839 (1.6288) | -20.789 (4.5189) | -5.668 (6.6271)
  GDS | -0.164 (0.4780) | -0.182 (0.1926) | 0.066 (0.4753) | -0.171 (0.3546) | 0.530 (0.5679) | -0.727 (0.8264)

6. Secondary Outcome: Correlation of Change in ADAS-Cog and SUVR
Description: Correlation between change from baseline to 36 month ADAS-Cog score and baseline global average SUVR by diagnostic group is provided below. ADAS-Cog scores (range 0-70) indicate performance on a series of 11 cognitive tasks where 0 indicates the highest level of cognitive performance and 70 indicates the lowest level of cognitive performance. Change in ADAS-Cog scores were calculated by subtracting the baseline score from the 36 month score (LOCF). A change in ADAS-Cog greater than 0 indicates a deterioration in cognitive performance whereas a change in ADAS-Cog less than 0 indicates improved cognitive performance. Standard Uptake Value Ratio (SUVR) is the ratio of tracer uptake in the cortex and cerebellum. SUVR values higher than 1 indicate greater amyloid burden in the cortex as compared to the cerebellum whereas scores less than 1 indicate the opposite.
Time Frame: Baseline and 36 months
Measure: Number; unit: Pearson Correlation Coefficient
Groups:
- Alzheimer's Disease: Subjects with a baseline clinical diagnosis of AD.
- Mild Cognitive Impairment: Subjects with a baseline clinical diagnosis of MCI.
- Cognitively Normal: Subjects with a baseline clinical diagnosis of CN.
Arm/Group | Alzheimer's Disease | Mild Cognitive Impairment | Cognitively Normal
Number analyzed (Participants) | 28 | 47 | 67
Pearson Correlation Coefficient | 0.364 | 0.502 | 0.308

ADVERSE EVENTS:
Description: The number of subjects at risk was determined by the number of subjects who received an injection of florbetapir F 18 at the 24 month time point of study 18F-AV-45-A11. As indicated in the participant flow group description, there were 36 MCI and 50 CN subjects who qualified for inclusion in the safety set.
Arm/Group | Alzheimer's Disease | Mild Cognitive Impairment | Cognitively Normal
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/36 | 0/50
Other Adverse Events (participants affected / at risk) | 0/0 | 1/36 | 1/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alzheimer's Disease (N=0) | Mild Cognitive Impairment (N=36) | Cognitively Normal (N=50)
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alzheimer's Disease (N=0) | Mild Cognitive Impairment (N=36) | Cognitively Normal (N=50)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less